CLINICAL TRIAL: NCT06214715
Title: Renal Resistive Index and Tissue Hypoperfusion Parameters and Prognosis Relationship in Septic Shock Patients
Brief Title: Renal Resistive Index in Septic Shock Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BVU-AR-MR-001
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Philips ultrasonography system — RRI will be measured by renal ultrasonography with a C5-1 convex probe using a Philips ultrasonography model device.

SUMMARY:
Septic shock is a condition of acute circulatory failure and is defined as a process that requires the use of vasopressors to ensure adequate tissue perfusion when hypotension develops. It is mainly characterized by abnormal peripheral vascular resistance; Therefore, improving vascular function and organ damage is crucial in the management of septic shock. Blood flow measurement with Doppler-based renal resistive index (RRI), which can be performed at the bedside, especially in renal abnormalities, is currently accepted as a tool to assess renal perfusion. With this simple, rapid and reproducible technique, the investigators determine RRI by evaluating systolic and diastolic blood velocity from Doppler flow waveforms in the intrarenal arcuate or interlobar arteries. Our aim is to investigate the relationship between renal resistive index (RRI) and global tissue hypoperfusion parameters and clinical outcomes in septic shock patients admitted to the intensive care unit and receiving invasive mechanical ventilator support.

DETAILED DESCRIPTION:
It is planned for patients who are admitted due to septic shock and need invasive mechanical ventilator support, who have a central venous catheter inserted for central venous pressure measurement and advanced monitoring, and who have undergone invasive arterial monitoring for close hemodynamic monitoring. After initial hemodynamic stabilization is achieved, RRI will be calculated by renal ultrasonography within 24 hours. Simultaneously with renal ultrasonography, blood samples will be taken from arterial and central venous catheters, partial arterial oxygen pressure (PaO2), partial arterial carbon dioxide pressure (PaCO2), partial central venous oxygen pressure (PcvO2) and partial central venous carbon dioxide pressure (PcvCO2), arterial Oxygen saturation (SaO2), central venous oxygen saturation (ScvO2), hemoglobin concentration and arterial lactate levels will be recorded. An attempt will be made to gain an idea about the course of the disease by comparing RRI with these global tissue hypoperfusion parameters.

ELIGIBILITY:
Inclusion Criteria:

* Followed up due to sepsis
* In need of intensive care follow-up
* In need of invasive mechanical ventilation
* Sofa score >2

Exclusion Criteria:

* Hypothermic patients (<35C)
* with chronic renal failure
* Pregnant women
* Those with renal artery stenosis
* Structural kidney damage
* Patient with previous renal surgery
* Intra-abdominal postoperative surgery patients
* Patients with atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is planned for patients who are admitted due to septic shock and need invasive mechanical ventilator support, who have a central venous catheter inserted for central venous pressure measurement and advanced monitoring, and who have undergone invasive arterial monitoring for close hemodynamic monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Renal resistive index | 24 hour
  The renal arterial resistive index (RI) is a sonographic index of intrarenal arteries defined as (peak systolic velocity - end-diastolic velocity) / peak systolic velocity. The normal range is 0.50-0.70

CONTACTS AND LOCATIONS:
Overall Officials: Monira Rahim, M.D., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No